CLINICAL TRIAL: NCT06339749
Title: Pregnancy Outcomes in Normotensive VS stage1 Hypertension: a Prospective Observational Study
Status: Recruiting | Type: Observational
Sponsor: FANG HE (Other)
Responsible Party: Sponsor-Investigator, FANG HE, Chief Physician/Professor of the Obstetrics Department, The Third Affiliated Hospital of Guangzhou Medical University
Organization: The Third Affiliated Hospital of Guangzhou Medical University (Other)
Other Study IDs: [2024] Ethics Review NO.040
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: stage1 Hypertension; Preeclampsia
Keywords: stage1 hypertension; Preeclampsia; observation; pregnancy outcomes
MeSH Terms: conditions — Pre-Eclampsia | interventions — Blood Pressure; Clinical Protocols

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Main study objective Groups: normotensive group: Main study objective Groups: normotensive group
  Interventions: Diagnostic Test: blood pressure
- Main study objective Groups: Stage 1 hypertension group: Main study objective Groups: Stage 1 hypertension group
  Interventions: Diagnostic Test: blood pressure
- Secondary objective grouping: Stage 1 hypertension low-risk group: Secondary objective grouping: Stage 1 hypertension low-risk group
  Interventions: Diagnostic Test: blood pressure; Other: Clinical protocols for preeclampsia risk screening
- Secondary objective grouping: Stage 1 hypertension high-risk group: Secondary objective grouping: Stage 1 hypertension high-risk group
  Interventions: Diagnostic Test: blood pressure; Other: Clinical protocols for preeclampsia risk screening

INTERVENTIONS:
Diagnostic Test: blood pressure — Based on first-trimester BP measurements, pregnant women were reclassified as normotensive (systolic BP < 120mmHg and diastolic BP <80mmHg on at least two occasions) and stage 1 hypertensive (systolic BP 130-139 mmHg and/or diastolic BP 80-89 mmHg on at least two occasions, without a diagnosis of chronic hypertension and/or elevated BP).
Other: Clinical protocols for preeclampsia risk screening — In this study, the risk factors of preeclampsia in pregnant women with combined maternal factors, MAP and PLGF were comprehensively analyzed by the "Bayesian rule" developed by the British Fetal Medicine Foundation (FMF). The online calculation website is: https://fetalmedicine.org/research/assess/preeclampsia/first-trimester.
  Groups: Secondary objective grouping: Stage 1 hypertension high-risk group; Secondary objective grouping: Stage 1 hypertension low-risk group

SUMMARY:
In 2017, the American College of Cardiology (ACC) and American Heart Association (AHA) guidelines built on evidence that elevated blood pressure increases cardiovascular mortality in the general population, Reclassification of BP; however, these diagnostic definitions do not include pregnant women, and whether newly diagnosed stage 1 hypertension affects pregnancy complications remains unclear. In this study, the combination of maternal factors, MAP and PLGF was used to comprehensively analyze the risk factors of preeclampsia through the "Bayesian rule" developed by the British Fetal Medicine Foundation (FMF). According to the guidelines and consensus, the pregnant women were considered to be at high risk when the calculated risk was higher than 1% of the population. To compare the pregnancy outcomes of women with normal blood pressure in the first trimester and stage 1 hypertension in different risk groups, and to find out whether screening for preeclampsia can be omitted for women with normal blood pressure in the first trimester, while screening for preeclampsia should still be performed for women with stage 1 hypertension as an independent moderate risk factor, and finally to optimize the screening strategy for preeclampsia.

DETAILED DESCRIPTION:
Based on first-trimester BP measurements, pregnant women were reclassified as normotensive (systolic BP < 120mmHg and diastolic BP <80mmHg on at least two occasions) and stage 1 hypertensive (systolic BP 130-139 mmHg and/or diastolic BP 80-89 mmHg on at least two occasions, without a diagnosis of chronic hypertension and/or elevated BP). At the same time, based on the 2019 FIGO pre-eclampsia screening guidelines, it is recommended that all pregnant women should be screened for pre-eclampsia in the first trimester. In this study, pregnant women who combined maternal factors, MAP and PLGF were analyzed by the "Bayesian rule" developed by the British Fetal Medicine Foundation (FMF). Its online computing website: https://fetalmedicine.org/research/assess/preeclampsia/first-trimester. The individual risk of preterm PE was calculated at 11-14+1 weeks of gestation using the British Fetal Medicine Foundation (FMF) algorithm. Previous risk was calculated based on maternal demographic characteristics and obstetric history. Therefore, 1/100 was selected as the cut-off value, ≥1/100 was registered as high risk of preeclampsia, < 1/100 was registered as low risk of preeclampsia. For people with high risk of preeclampsia (≥1/100) evaluated in the first trimester, low-dose aspirin prevention for preeclampsia is recommended between 12 and 28 weeks of gestation (preferably before 16 weeks). And continued until 36 weeks. To compare the pregnancy outcomes of women with normal blood pressure in the first trimester and stage 1 hypertension in different risk groups, and to find out whether screening for preeclampsia can be omitted for women with normal blood pressure in the first trimester, while screening for preeclampsia should still be performed for women with stage 1 hypertension as an independent moderate risk factor, and finally to optimize the screening strategy for preeclampsia.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old;
2. single live fetus with normal NT at 11-14+1 weeks of gestation;
3. Blood pressure < 140/90 mmHg before 14+1 week of gestation;
4. Plan to have prenatal examination and delivery in our hospital;
5. Sign informed consent.

Exclusion Criteria:

Underlying diseases (chronic hypertension, type 1 or type 2 diabetes, kidney disease, autoimmune disease).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All the subjects were pregnant women who delivered in our hospital.
Sampling Method: Probability Sample
Enrollment: 626 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
preeclampsia | After 20 weeks of gestation until the end of delivery
  The criteria for preeclampsia were based on the Chinese Guidelines for the Diagnosis and Treatment of Hypertensive Disorders in Pregnancy, which were systolic blood pressure ≥140mmHg and/or diastolic blood pressure ≥90mmHg after 20 weeks of gestation, accompanied by any one of the following: Urine protein ≥0.3 g/24h, or urine protein/creatinine ratio ≥0.3, or random urine protein ≥ (+). There is no proteinuria, but there is involvement of any of the following organs or systems: important organs such as the heart, lungs, liver, kidney, or abnormal changes in the blood system, digestive system, nervous system, placental-fetal involvement.

SECONDARY OUTCOMES:
Preterm birth | After 20 weeks of gestation until the end of delivery
  Preterm birth were defined as live birth with gestational age < 37 weeks.
fetal intrauterine growth restriction (FGR) | After 20 weeks of gestation until the end of delivery
  FGR is a condition in which fetal growth does not reach its genetic potential due to the influence of maternal, fetal, placental and other pathological factors, mostly manifested as fetal ultrasonographic estimated weight or abdominal circumference below the 10th percentile for gestational age.
Severe complications of preeclampsia | After 20 weeks of gestation until the end of delivery
  hemolysis，elevated liver enzymes and low platelets count syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Fang He, M.D, Principal Investigator — The Third Affiliated Hospital of Guangzhou Medical University
Locations (1):
- FANG HE, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No